CLINICAL TRIAL: NCT04571372
Title: Prognostic Value of Soluble Urokinase-type Plasminogen Activator Receptor in Valvular Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-0620
Record Dates: First submitted 2020-08-13; First posted 2020-10-01 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Severe Aortic Stenosis or Severe Aortic Regurgitation
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with severe aortic stenosis or severe aortic regurgitation: Patients with severe aortic stenosis or severe aortic regurgitation

SUMMARY:
This study investigates the association between level of suPAR and valvular heart disease in patients who have severe aortic stenosis or severe aortic regurgitation using commercially available suPARnostic standard enzyme-linked immunosorbent assay (ViroGates, Denmark)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 yrs
* Severe aortic stenosis or severe aortic regurgitation
* Agree to consent for self
* Can follow-up for the next 2 years

Exclusion Criteria:

* Pre-existing acute kidney injury
* Pre-existing end stage kidney disease: estimated glomerular filtration rate (eGFR) ≤15 ml/min/1.73m2 or receiving renal replacement therapy
* On ECMO or IABP
* Life expectancy < 12 months
* Pregnancy

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe aortic stenosis or severe aortic regurgitation
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse clinical outcomes | Immediate post operation
  Composite of all-cause death, cardiovascular mortality, and worsening of kidney function
Number of participants with adverse clinical outcomes | 2 years after recruiting
  Composite of all-cause death, cardiovascular mortality, and worsening of kidney function

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koller L, Stojkovic S, Richter B, Sulzgruber P, Potolidis C, Liebhart F, Mortl D, Berger R, Goliasch G, Wojta J, Hulsmann M, Niessner A. Soluble Urokinase-Type Plasminogen Activator Receptor Improves Risk Prediction in Patients With Chronic Heart Failure. JACC Heart Fail. 2017 Apr;5(4):268-277. doi: 10.1016/j.jchf.2016.12.008. PMID 28359415
- [Background] Hayek SS, Sever S, Ko YA, Trachtman H, Awad M, Wadhwani S, Altintas MM, Wei C, Hotton AL, French AL, Sperling LS, Lerakis S, Quyyumi AA, Reiser J. Soluble Urokinase Receptor and Chronic Kidney Disease. N Engl J Med. 2015 Nov 12;373(20):1916-25. doi: 10.1056/NEJMoa1506362. Epub 2015 Nov 5. PMID 26539835
- [Background] Hayek SS, Leaf DE, Samman Tahhan A, Raad M, Sharma S, Waikar SS, Sever S, Camacho A, Wang X, Dande RR, Ibrahim NE, Baron RM, Altintas MM, Wei C, Sheikh-Hamad D, Pan JS, Holliday MW Jr, Januzzi JL, Weisbord SD, Quyyumi AA, Reiser J. Soluble Urokinase Receptor and Acute Kidney Injury. N Engl J Med. 2020 Jan 30;382(5):416-426. doi: 10.1056/NEJMoa1911481. PMID 31995687